CLINICAL TRIAL: NCT02890277
Title: Treatment of Nonneoplastic Epithelial Disorders of Skin and Mucosa of Vulva With High Intensity Focused Ultrasound
Brief Title: Nonneoplastic Epithelial Disorders of Vulva and High Intensity Focused Ultrasound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinan Military General Hospital (Other)
Responsible Party: Principal Investigator, Geping Yin, Professor/Surgeon,Leader of Department of Gynecology, Jinan Military General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JNJQ201408
Record Dates: First submitted 2015-02-14; First posted 2016-09-07 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Vulva Intraepithelial Nonneoplastic
MeSH Terms: interventions — formaldehyde, meta-cresolsulfonic acid drug combination

ARMS (1):
- Treatment group (Experimental)
  Interventions: Device: the high intensity focused ultrasound (Mianyang Sonic electronic LLC); Drug: Fu Tiankang disposable vaginal filling suppository, Albothyl (Policresulen Solution) , and the gynecologic medical antimicrobial dressing gel (chitosan gel).

INTERVENTIONS:
Device: the high intensity focused ultrasound (Mianyang Sonic electronic LLC)
Drug: Fu Tiankang disposable vaginal filling suppository, Albothyl (Policresulen Solution) , and the gynecologic medical antimicrobial dressing gel (chitosan gel).

SUMMARY:
Nonneoplastic epithelial disorders of skin and mucosa of vulva refer to a group of chronic diseases shown as female genital skin and mucosal tissue degeneration and pigmentation change. The main symptoms are vulval itching, squamous cell hyperplasia, vulval and perianal skin atrophy or thinning, hypopigmentation. The current treatments are primarily local drug or surgical treatments. However, the effect is not good enough, but the diseases often recur and severely affect patients' quality of life. In this study, the investigators combined the technology of high intensity focused ultrasound (HIFU) (ultrasound device made by Mianyang Sonic electronic LLC, Mianyang China, registration number: 2005-2230099} with special drug to treat. The data from colposcopy and biopsy pathology were collected before and after treatment to create the objective identifying degree of the disease by with "grading methods" and evaluate the treatment effect. At the meantime, the standardized treatment procedure, methods and efficacy criterion were all stipulated to achieve satisfactory results, which could be used to clinical treatments. So far, the investigators have not seen similar study reported internationally.

ELIGIBILITY:
Inclusion criteria:

* patients with clinically and biopsy confirmed non-neoplastic lesions of genital skin and mucous membrane (non-neoplasia epithelial disorders of skin and mucosa of vulva).

Symptoms include repeated itching, discoloration, rhagades, loss of skin elasticity and dyspareunia that affect the patients' quality of life.

Exclusion criteria:

* atypical hyperplasia or vulvar cancer confirmed by biopsy of genital lesions;
* vulvovaginal or other gynecological trauma, acute inflammatory diseases and other acute illness in need of urgent care;
* combined with other serious gynecological diseases (symptomatic hysteromyoma, ovarian tumor, etc.), and/or severe organ diseases (such as heart, lung, brain and renal disease/failure) that need immediate treatment;
* other type of cancers that require urgent care.

Ages: 18 Years to 78 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Grading changes of nonneoplastic epithelial disorders from colposcopy and biopsy pathology | One month before treatment and 2,4,6 weeks and 2,6,12,24 monthes after treatment
  The data from colposcopy and biopsy pathology were collected before and after treatment to create the objective identifying degree of the disease by with "grading methods" and evaluate the treatment effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinan Military General Hospital, Jinan, Shandong, China